CLINICAL TRIAL: NCT06782893
Title: COUGH-LESS: Chronic COUGH Management in Interstitial Lung DisEase - Non-pharmacological Strategies and Solutions
Brief Title: Chronic COUGH Management in Interstitial Lung DisEase
Acronym: COUGH-LESS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other); Centro Hospitalar do Baixo Vouga (Other); Centro Hospitalar de Entre o Douro e Vouga (Other)
Responsible Party: Principal Investigator, Prof Ana Oliveira, Assistant professor, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023.01387.BDANA
Record Dates: First submitted 2024-07-30; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-07

CONDITIONS: Interstitial Lung Disease; Chronic Cough
Keywords: Chronic Cough; Interstitial Lung Disease; Non-pharmacological cough control therapy
MeSH Terms: conditions — Lung Diseases, Interstitial; Chronic Cough

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- COUGH-LESS Programme (Experimental)
  Interventions: Behavioral: Non-pharmacological cough control therapy
- Control Group (Sham Comparator)
  Interventions: Behavioral: Healthy lifestyle

INTERVENTIONS:
Behavioral: Non-pharmacological cough control therapy — Over seven weeks (1 session per week, except session 5, which will be 2 weeks after session 4) using a one-on-one hybrid model. In session 1, participants will receive general education about chronic cough, introduction to cough suppression and goal setting. Session 2 will cover education about chronic cough in ILD, cough triggers and training in cough suppression techniques. Session 3 will focus on hydration techniques, laryngeal hygiene, and breathing exercises to control coughing. Session 4 will reinforce all aspects of non-pharmacological cough control treatment, and session 5 will explore the sustainability of cough control strategies after the program using real-life case scenarios.
  Arms: COUGH-LESS Programme
Behavioral: Healthy lifestyle — Over seven weeks (1 session per week, except session 5, which will be 2 weeks after session 4) using a one-on-one hybrid model. In session 1, participants will receive general education about exercise and physical activity. Session 2 will cover education about diet. Session 3 will focus on stress management. Session 4 will cover relaxation techniques, and session 5 will reinforce all aspects previously considered.
  Arms: Control Group

SUMMARY:
Interstitial Lung Disease (ILD) includes chronic, disabling and progressive respiratory conditions marked by lung inflammation and fibrosis. The quality of life and functionality of people with ILD is affected by a plethora of debilitating symptoms such as dyspnoea fatigue and cough. Among them, chronic cough (a cough lasting more than 8 weeks) reigns as one of the most prevalent and challenging, despite receiving far less attention from researchers than other symptoms. Chronic cough affects up to 8 out of 10 individuals with ILD and it is associated with a worse prognosis, mortality, and the need for lung transplantation. This condition showed a significant impact in people's life (e.g., urinary incontinence, speech interferences, depression, chest pain, couples sleeping in separate bedrooms, avoidance of public areas, reduced social interaction, and work absenteeism), further contributing to the decreased health-related quality of life experienced by this population. Managing chronic cough is, therefore, urgently needed. The general aim of this study is to explore the effects of a non-pharmacological cough control treatment on cough-related quality of life in people with ILD. The specific aims of this study are: i) to explore short- and mid-term effects of the non-pharmacological cough control treatment on cough related outcomes (e.g., cough frequency and intensity, dyspnoea, fatigue, cough self-efficacy, health-related quality of life and emotional status); ii) to identify (if any) adverse effects of this therapy.

DETAILED DESCRIPTION:
Interstitial Lung Disease (ILD) comprises chronic, disabling, and progressive respiratory conditions marked by lung inflammation and fibrosis. The quality of life and functionality of people with ILD is affected by a plethora of debilitating symptoms such as dyspnoea, fatigue, and cough. Among them, chronic cough reigns as one of the most prevalent and challenging, despite receiving far less attention from researchers than other symptoms.

Chronic cough (a cough lasting for > 8 weeks) and affects up to 8 out of 10 individuals with ILD. It is associated with a worse prognosis, mortality, and the need for lung transplantation. This condition also causes urinary incontinence, interferes with speech, and presents psychosocial and physical manifestations, such as depression and chest pain. Chronic cough can also lead to relationship problems, such as couples sleeping in separate bedrooms, avoidance of public areas, reduced social interaction, and work absenteeism, further contributing to the decreased health-related quality of life experienced by this population. Managing chronic cough is, therefore, urgently needed.

Currently, there is no approved drug to manage chronic cough in people with ILD. Conversely, non-pharmacologic cough control therapies have demonstrated similar efficacy without side effects. Studies have shown that non-pharmacological cough control therapy can improve cough-related quality of life and reduce cough frequency in individuals with refractory (i.e., cough that lasts despite optimal treatment) chronic cough. Promising results were observed in a case-study on people with chronic cough and ILD. However, well-designed randomized controlled trials (RCTs) with adequate power are needed to establish the effects of non-pharmacological cough control therapy on people with ILD.

The primary aim of this study is to explore the effects of a non-pharmacological cough control treatment on cough-related quality of life in people with ILD. The specific aims of this study are: i) to explore short- and mid-term effects of the non-pharmacological cough control treatment on cough related outcomes (e.g., cough frequency and intensity, dyspnea, fatigue, cough self-efficacy, health-related quality of life and emotional status); ii) to identify (if any) adverse effects of this therapy.

COUGH-LESS randomized trial Potential participants will be identified and recruited through the pulmonology services of the Centro Hospitalar do Baixo Vouga (CHBV) and Centro Hospitalar de Entre-o-Douro e Vouga (CHEDV).

Study design Participants will be randomly assigned to an experimental (EG) or control group (CG) using an online software. Assessments will be conducted at baseline, post-intervention and 3 and 6 months after the intervention. To detect a 2-point between-group difference in the LCQ after 5 weeks, 20 participants per group (n=40) will be required, with 80% power and a significance level of 5%. Previous studies indicate losses to follow up of 50% and thus we will aim to recruit 60 individuals.

Data collection Assessments will be conducted at baseline, post-intervention and 3 and 6 months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

i) Adults (>18 years old) ii) Clinical diagnosis of ILD iii) Presenting chronic cough (> 8 weeks of duration) iv) People with access to a virtual meeting platform/telephone.

Exclusion Criteria:

i) Self-reports of moderate or large sputum production (> 2 tablespoons); ii) Actual or suspected exacerbation of the respiratory condition in the last month; iii) Upper respiratory tract infection (e.g. cold); iv) Use of angiotensin-converting enzyme inhibitor medication; v) Changes in prescribed medication in the last month; vi) Signs of cognitive impairment or significant cardiovascular, neurological and/or musculoskeletal disease that may limit participation in the program; vii) Inability to read or speak Portuguese; viii) Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2027-12-20 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in Leicester Cough Questionnaire (LCQ) | One measurement will be assessed at baseline, 7 weeks after interventions and 3 and 6 months after the intervention.
  The LCQ is a reliable, responsive questionnaire recommended by various guidelines for assessing chronic cough. This questionnaire comprises 21 questions referring to the two weeks prior to completing it. The LCQ assesses three domains (psychological, social and physical) and also gives a total score. The maximum score that can be obtained on the LCQ is 21 points in total (7 in each domain) where higher scores translate into a higher quality of life related to coughing.

SECONDARY OUTCOMES:
Change in Modified British Medical Research Council Dyspnea Scale (mMRC) | One measurement will be assessed at baseline, 7 weeks after interventions and 3 and 6 months after the intervention.
  The mMRC has been validated for the Portuguese population and is a predictor of increased severity in people with ILD.
Change in Cough Visual Analogic Scale (CVAS) | One measurement will be assessed at baseline, 7 weeks after (post-intervention) and 3 and 6 months after the intervention.
  The CVAS will be used to measure intensity and frequency of cough. This scale consists of a 10 cm line ranging from 0 (no severity/intensity) to 10 (extreme severity/intensity) and is moderately responsive.
Change in Chronic Airways Assessment Test (CAAT) | One measurement will be assessed at baseline, 7 weeks after (post-intervention) and 3 and 6 months after the intervention.
  CAT will be used to measure quality of life related to respiratory symptoms. This scale ranges from 0 to 45, where higher values mean a lower quality of life related to respiratory symptoms in people with ILD.
Change in One minute sit-to-stand test (1min-STS) | One measurement will be assessed at baseline, 7 weeks after (post-intervention) and 3 and 6 months after the intervention.
  The 1min-STS will be used to assess functional capacity. It will be counted the maximum number of repetitions completed in 1 minute while sitting and standing on a chair.
Six-minute Walking Test (6MWT) | One measurement will be assessed at baseline, 7 weeks after (post-intervention) and 3 and 6 months after the intervention.
  The 6MWT will be used also to measure functional capacity and has been validated in people with ILD. The walked total distance during the six minutes will be counted.
Change in Cough Hypersensitivity Questionnaire (CHQ) | One measurement will be assessed at baseline, 7 weeks after (post-intervention) and 3 and 6 months after the intervention.
  The CHQ comprises 23 questions related to cough-causing stimuli and coughing sensations. This questionnaire scores rages from 0 to 23 points, where higher scores mean a greater presence and severity of stimuli and triggers of cough and sensations in the larynx.
Change in Hospital Anxiety and Depression Scale (HADS) | One measurement will be assessed at baseline, 7 weeks after (post-intervention) and 3 and 6 months after the intervention.
  HADS is an easy-to-use scale that is subdivided into two domains (anxiety symptoms and depressive symptoms). Their score varies from 0 to 21 in each subdomain, where a score between 0 and 7 is considered 'normal', between 8 and 10 indicates a "mild" level, between 11 and 14 a "moderate" level, and between 15 and 21 "severe" levels of anxiety and depression symptoms.
Change in Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-FS) | One measurement will be assessed at baseline, 7 weeks after (post-intervention) and 3 and 6 months after the intervention.
  FACIT-FS assesses fatigue where a higher score translates into lower fatigue. This scale is commonly used in the ILD population to assess fatigue, presenting good reliability and feasibility.
Change in King's Brief Interstitial Lung Disease (K-BILD) | One measurement will be assessed at baseline, 7 weeks after (post-intervention) and 3 and 6 months after the intervention.
  K-BILD will be used to assess health related quality of life. This scale encompasses three domains: psychological, dyspnoea, activities, and respiratory symptoms where higher scores define a high health related quality of life.
Interviews | One measurement will be assessed at baseline and 7 weeks after (post-intervention)
  Participants will be invited to take part in face-to-face, semi-structured individual interviews the impact of both interventions (control and experimental group).
Adherence to the COUGH-LESS programme | Only one measurement will be assessed after 7 weeks after baseline (post-intervention).
  Participants' number of sessions attended to the intervention will be registered.
Occurrence of adverse events | One measurement will be assessed at 7 weeks after baseline (post-intervention) and 3 and 6 months after the intervention.
  The occurrence of adverse events in participants will be registered according to CTCAE v4.0.

OTHER OUTCOMES:
Change in number of hospitalizations | One measurement will be assessed at 7 weeks after baseline (post-intervention) and 3 and 6 months after the intervention.
  Patients' number of hospitalizations in the previous year and during the follow-up period, as well as the length of stay for each hospitalization, will be assessed by asking the patient to self-report.
Change in acute exacerbations | One measurement will be assessed at 7 weeks after baseline (post-intervention) and 3 and 6 months after the intervention.
  Patients' number of acute exacerbations will be assessed by asking the patient to self-report.
Interstitial Lung Disease- Gender, Age and Physiology model (ILD-GAP model) | Only one measurement will be assessed on baseline. This will be used as a descriptive measure.
  ILD-GAP model measures the severity of the disease based on the diagnosis, sex and respiratory function test values to create a score that can vary between 0 and 8. The greater the severity of the disease, the higher the ILD-GAP model.

CONTACTS AND LOCATIONS:
Locations (1):
- Aveiro University, Aveiro, Portugal

IPD SHARING:
Plan to Share IPD: No